CLINICAL TRIAL: NCT06376045
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose Ranging Study to Assess the Efficacy and Safety of Rocatinlimab in Adult Subjects With Moderate-to-severe Asthma
Brief Title: A Phase 2, Dose Ranging Study Assessing Rocatinlimab in Moderate-to-severe Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220093
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Moderate to severe asthma; Rocatinlimab; AMG 451; KHK4083
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Arm A: Placebo (Placebo Comparator): Participants will receive placebo by subcutaneous (SC) injection during the blinded treatment period.
  Interventions: Drug: Placebo
- Treatment Arm B: Dose 1 Rocatinlimab (Experimental): Participants will receive dose 1 rocatinlimab by SC injection during the blinded treatment period.
  Interventions: Drug: Rocatinlimab
- Treatment Arm C: Dose 2 Rocatinlimab (Experimental): Participants will receive dose 2 rocatinlimab by SC injection during the blinded treatment period.
  Interventions: Drug: Rocatinlimab
- Treatment Arm D: Dose 3 Rocatinlimab (Experimental): Participants will receive dose 3 rocatinlimab by SC injection during the blinded treatment period.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Rocatinlimab will be administered by SC injection.
  Other Names: AMG 451
  Arms: Treatment Arm B: Dose 1 Rocatinlimab; Treatment Arm C: Dose 2 Rocatinlimab; Treatment Arm D: Dose 3 Rocatinlimab
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Treatment Arm A: Placebo

SUMMARY:
The primary objective of this study is to describe the efficacy of rocatinlimab in reducing asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 and 75.
* Asthma diagnosed by a physician for ≥ 12 months prior to the screening visit.
* Existing therapy with medium-dose to high doses of inhaled corticosteroids (ICS) (defined as > 250 µg fluticasone propionate or equivalent ICS) in combination with at least 1 additional controller medication (eg, LABA, leukotriene receptor antagonist [LTRA], LAMA, methylxanthine, oral corticosteroids up to a daily dose of 10 mg prednisone equivalent) for at least 90 days prior to the screening visit with a stable dose for at least 30 days prior to the screening visit.
* Documented history of ≥ 1 asthma exacerbation in the past year prior to the screening visit, with at least 1 exacerbation during treatment with medium-dose to high doses of ICS (> 250 μg fluticasone propionate or equivalent ICS).
* Morning pre-BD FEV1 ≥ 35% and ≤ 90% of predicted normal at the screening visit and day 1 pre-randomization visits.
* ACQ-6 score ≥ 1.5 at the day 1 pre randomization visit.

Exclusion Criteria:

* Asthma exacerbation that results in emergency treatment or hospitalization, or treatment with systemic steroids at any time from 30 days prior to the day 1 pre randomization visit.
* Any clinically important pulmonary disease other than asthma.
* Current smoker, including active vaping of any products and/or marijuana, or former smoker with cessation within 6 months of screening, or history of > 10 pack-years.
* Suspicion of, or confirmed, coronavirus disease 2019 (COVID-19) infection during the screening period including known history of COVID-19 infection within 4 weeks prior to Screening; mechanical ventilation or extracorporeal membrane oxygenation (ECMO) secondary to COVID-19 within 3 months prior to screening; participants with COVID-19 infection who have not yet sufficiently recovered to participate in the procedures of a clinical trial.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antiviral, antiparasitic, antiprotozoal, or antifungals which has not completely resolved, or for which therapy has not been completed, within 4 weeks before day 1 pre-randomization visit.
* Positive or indeterminate QuantiFERON GOLD from central laboratory at screening.
* Active malignancy; multiple myeloma; myeloproliferative or lymphoproliferative disorder; or a history of any of these conditions within 5 years prior to informed consent
* History of major immunologic reaction to any other biologic product or any excipient of rocatinlimab.
* Diagnosis of a helminth parasitic infection within 6 months prior to day 1 pre-randomization visit that had not been treated with or had failed to respond to standard of care therapy.
* Evidence of human immunodeficiency virus (HIV) infection or positive for HIV antibodies at screening or current acquired, common variable or inherited, primary or secondary immunodeficiency.
* Active and non-virally suppressed hepatitis B infection at initial screening,
* Positive for hepatitis C virus (HCV) antibody at screening with confirmed positive HCV RNA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of Composite Endpoint for Exacerbations (CompEx) Events During the Blinded Treatment Period | Up to Week 48

SECONDARY OUTCOMES:
Annualized Asthma Exacerbation Rate (AAER) | Up to Week 48
Change From Baseline in Pre-bronchodilator (BD) Forced Expiratory Volume in 1 Second (FEV1) | Baseline and Week 48
Change From Baseline in Asthma Control Questionnaire 6 (ACQ-6) Score at Week 48 | Baseline and Week 48
Change From Baseline in Pre-BD FEV1 | Up to 62 weeks
Change From Baseline in Asthma Symptom Diary (ASD) Score | Up to Week 48
Number of Participant Achieving ACQ-6 Response at Week 48 | Week 48
Change From Baseline in ACQ-6 | Up to Week 48
Change From Baseline in Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ [S]) Self-Administered Score | Baseline, Weeks 12, 24, 36 and 48
Number of Participants Achieving AQLQ (S) Response at Week 48 | Up to Week 48
Annualized Rate of Asthma Exacerbation Leading to Hospitalization or Emergency Room Visits During the Blinded Treatment Period | Up to Week 48
Time to First Asthma Exacerbation Event | Up to 62 weeks
Time to First CompEx Event | Up to 62 weeks
Number of Participants with a CompEx Event During the Double Blinded Treatment Period | Up to Week 48
Annualized Rate of CompEx Events | Weeks 12, 24 and 36
Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) Levels | Up to 62 weeks
Serum Rocatinlimab Concentrations | Up to 62 weeks
Trough Concentration (Ctrough) of Rocatinlimab | Up to 62 weeks
Number of Participants with Treatment-emergent Adverse Events | Up to 62 weeks
Number of Participants with Serious Adverse Events | Up to 62 weeks
Number of Participants with Anti-rocatinlimab Antibody Formation | Up to 62 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (154):
- United States (48):
  - Kern Research Inc, Bakersfield, California
  - Orso Health Inc, La Jolla, California
  - Imax Clinical Trials, La Palma, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Downtown Los Angeles Research Center, Inc, Los Angeles, California
  - NewportNativeMD, Inc, Newport Beach, California
  - University of California Irvine, Orange, California
  - Apex Clinical Research, San Diego, California
  - Allergy and Asthma Clinical Research, Walnut Creek, California
  - Allianz Research Institute Westminster, Westminster, California
  - St Francis Medical Institute, Clearwater, Florida
  - BioMed Research Institute, Miami, Florida
  - Bright Research Center LLC, Miami, Florida
  - Infinity Life Research Group, Tamarac, Florida
  - Clinical Research Trials of Florida Inc, Tampa, Florida
  - AllerVie Clinical Research- Columbus, Columbus, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Sneeze, Wheeze, and Itch Associates, LLC, Normal, Illinois
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Chesapeake Clinical Research Inc, White Marsh, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Respiratory Medicine Research Institute of Michigan, plc, Ypsilanti, Michigan
  - Midwest Chest Consultants, PC, Saint Charles, Missouri
  - Montana Medical Research, Missoula, Montana
  - Somnos Clinical Research, Lincoln, Nebraska
  - Hudson County Clinical Trials Research Center, Union City, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Duke Asthma Research Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center LLC, Cincinnati, Ohio
  - OK Clinical Research, Edmond, Oklahoma
  - Velocity Clinical Research Medford, Medford, Oregon
  - Clinical Research Associates of Central Pennsylvania, DuBois, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Allergy Asthma and Sinus Center, Knoxville, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - TTS Research, Boerne, Texas
  - TEN20 Clinical Research, Carrollton, Texas
  - Alina Clinical Trials, LLC, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Ace Proactive, Plano, Texas
  - South Texas Allergy and Asthma Medical Professionals, San Antonio, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Pioneer Research Solutions Inc, Sugar Land, Texas
- Argentina (10):
  - Fundacion Respirar - Centro Medico Dra De Salvo, CABA, Buenos Aires
  - Centro de Osteopatias Medicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Enfisema para el Estudio y Tratamiento de las Enfermedades Cronicas del Aparato Respirador, Mar del Plata, Buenos Aires
  - Ierim Instituto de Enfermedades Respiratorias e Investigacion Clinica, San Juan Bautista, Buenos Aires
  - InAER - Investigaciones en Alergia y Enfermedades Respiratorias, Buenos Aires, Distrito Federal
  - Fundacion Grupo Colaborativo Rosario Investigacion y Prevencion medica, Rosario, Santa Fe Province
  - Centro Integral de Medicina Respiratoria, San Miguel de Tucumán, Tucumán Province
  - Cemer Centro Medico de Enfermedades Respiratorias, Florida, Vicente Lopez
  - Instituto Medico Insares SA, Mendoza
  - Fundacion Scherbovsky, Mendoza
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Bulgaria (5):
  - Medical Center Pulmo - 2018 EOOD, Haskovo
  - Specialized Hospital for Active Treatment of Pneumo-phthisiatric Diseases Dr Dimitar Gramatikov, Rousse
  - Medical Center Excelsior OOD, Sofia
  - Diagnostic-Consultative Center Convex OOD, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora
- Canada (5):
  - University of Calgary - Cumming School of Medicine, Calgary, Alberta
  - Centre for Lung Health, Vancouver, British Columbia
  - St Pauls Hospital Pacific Lung Health Centre, Vancouver, British Columbia
  - Dynamic Drug Advancement Limited, Ajax, Ontario
  - Kanata Allergy Clinic, Ottawa, Ontario
- Chile (5):
  - Centro de Investigacion Curico, Curicó
  - Sociedad Medica SyG Limitada, Santiago
  - Centro De Investigaciones Medicas Respiratorias, Santiago
  - Icegclinic, Santiago
  - Centro de Investigacion del Maule, Talca
- China (16):
  - Hefei First Peoples Hospital, Hefei, Anhui
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Peoples Hospital of Huizhou, Huizhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Changsha Central Hospital, Changsha, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Jiangxi Provincial Peoples Hospital, Nanchang, Jiangxi
  - Pingxiang Peoples Hospital, Pingxiang, Jiangxi
  - Heze Municipal Hospital, Heze, Shandong
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
- Colombia (3):
  - Corporacion Hospitalaria Juan Ciudad, Mederi, Bogota, Cundinamarca
  - Solano y Terront Servicios Medicos SAS - Unidad Integral de Endocrinologia Uniendo, Bogota, Cundinamarca
  - Mediservis del Tolima IPS SAS, Ibagué, Tolima Department
- Czechia (4):
  - MUDr I Cierna Peterova sro, Brandýs nad Labem-Stará Boleslav
  - Meditrial sro, Jindřichův Hradec
  - MUDr Josef Veverka, Rokycany
  - Kasmed sro, Tábor
- Hong Kong (3):
  - Hong Kong Center for Clinical Research, Hong Kong
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Hungary (4):
  - Edelenyi Koch Robert Korhaz es Rendelointezet, Edelény
  - Erzsebet Gondozohaz, Gödöllő
  - Puspokladanyi Egeszsegugyi Szolgaltato Intezmeny, Püspökladány
  - Allergo-Fot Kft, Százhalombatta
- Japan (12):
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Medical corporation Syureikai Tohno Chuo Clinic, Mizunami-shi, Gifu
  - Idaimae Minami Yojo Naika Clinic, Sapporo, Hokkaido
  - Sakaide City Hospital, Sakaide-shi, Kagawa-ken
  - Kamei Internal medicine and Respiratory Clinic, Takamatsu, Kagawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi, Osaka
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Tokyo Shinagawa Hospital Social Medical Corporation Association Tokyokyojuno-kai, Shinagawa-ku, Tokyo
- Mexico (4):
  - Centro de investigacion medico biologica y terapia avanzada, Guadalajara, Jalisco
  - cicum San Miguel, Guadalaja, Jalisco
  - Icaro Investigaciones en Medicina, Chihuahua City
  - Unidad de Investigacion cima, Chihuahua City
- Poland (8):
  - Centrum Medycyny Oddechowej Mroz Spolka Jawna, Bialystok
  - Klimed Marek Klimkiewicz, Bychawa
  - GynCentrum Sp zoo NZOZ Holsamed, Katowice
  - Centrum Medyczne All-Med Badania kliniczne, Krakow
  - Diamond Clinic Spolka z Ograniczona Odpowiedzialnoscia Diamond Medical Center, Krakow
  - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olech-Cudzik Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Ewa Springer Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej, Poznan
  - Centrum Badan Klinicznych Piotr Napora lekarze spolka partnerska, Wroclaw
- Romania (5):
  - Spitalul de Pneumoftiziologie Bacau, Bacau
  - Spitalul de Pneumoftiziologie Leon Daniello, Cluj-Napoca
  - Spitalul Clinic de Boli Infecțioase si Pneumoftiziologie Victor Babes Craiova, Craiova
  - Medical Center, Deva
  - Spitalul Judetean de Urgenta Sf Ioan cel Nou Suceava, Suceava
- South Korea (8):
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Eunpyeong St Marys Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Veterans General Hospital - Taichung, Taichung
  - Taipei Medical University Hospital, Taipei
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla
- United Kingdom (5):
  - Lakeside Healthcare, Corby
  - CPS Research, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - 4 Medical Clinical Solutions, Manchester
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com